CLINICAL TRIAL: NCT00425516
Title: Clinical Trial of the Neoadjuvant Standard Chemotherapy 3 FEC 100 + 3 TAXOTERE Protocol Versus the Same Protocol Adapted as a Function of Clinical Response
Brief Title: Breast Cancer Treated by Neoadjuvant Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJP AU651/Afssaps060744
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2007-02

CONDITIONS: Individualized Chemotherapy
Keywords: neoadjuvant chemotherapy; breast cancer; sequential treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Fluorouracil; Epirubicin; Cyclophosphamide

ARMS (2):
- standard (A) (No Intervention): 3 FEC100 followed 3 Taxotere
- Modulated (B) (Experimental): possibility treatments receive: 2 FEC100 followed by 4 Taxotere 4 FEC100 followed by 2 Taxotere 6 FEC 100
  Interventions: Drug: Taxotere; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Taxotere
  Other Names: Docetaxel
  Arms: Modulated (B)
Drug: 5-Fluorouracil
  Arms: Modulated (B)
Drug: Epirubicin
  Arms: Modulated (B)
Drug: Cyclophosphamide
  Arms: Modulated (B)

SUMMARY:
Neoadjuvant chemotherapy, known as "first" or "induction chemotherapy" in the therapeutic assumption of breast cancer is based on the narrow dependence preclinically revealed between primary tumour, tumoral angiogenesis and growth of distant metastases.

The results of the Aberdeen Group (Smith et al, 2002 ; Hutcheon et al, 2003), of the NSABP B27 trial (Bear et al, 2003) and of the Gepar-Duo Group (Von Minckwitz et al, 2002) have shown that a sequential protocol, using docetaxel after an anthracycline-based combination, allowed a better clinical response leading to more frequent conservative surgeries and, more importantly, to an increase in the rate of complete pathological response, assessing a better efficacy.

The use of a reference adjuvant protocol as a neo-adjuvant treatment is fully admissible because 7 randomized trials have shown a perfect equivalence between an adjuvant protocol and the same chemotherapy given as an induction treatment Even keeping the principle of a sequential treatment, a crucial question is to know if this sequential treatment should be the same for all patients, or if the oncologist could get a better complete pathological response, disease-free or overall survival rates by an adaptation of treatment to the objective result beginning after 2 FEC 100 courses by modulation of the following courses.

We will use as a primary regimen 3 FEC cycles + 3 TAXOTERE cycles, a standard adjuvant regimen (noted in the Temporary Protocol of Treatment of the Inca page 5 (October 2005) as well as in Saint Paul de Vence 2005 recommendations for adjuvant chemotherapy (Oncologie -- volume 7 - N°5, August 2005, p 370). This standard treatment will be compared to the same chemotherapy modulated in its repartition according to results obtained by subsequent tumor evaluations during induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histological proof of non metastatic breast cancer, whose clinical tumor diameter is > 2 cm, or < 2 cm, but situated in areolar area of the nipple.
* T2-T3, N0-N1 tumor, non-inflammatory, unilateral, non-metastatic, grade II - III, HER2-neu negative, without extension beyond the breast and axillar area.
* Performance Status = 0-1 WHO.
* Patient non pretreated for breast cancer.
* Patient without cardiac pathology and without anthracyclines contra-indication (assessed by normal ejection fraction).
* Normal haematological, renal and hepatic functions : PNN > 2.109 /l, platelets > 100. 109 /l, Hb > 10 g/dl, normal bilirubin serum , ASAT and ALAT < 2,5 ULN, alkaline phosphatases < 2,5 ULN, creatinin < 140 µmol/l or creatinin clearance > 60 ml/min
* Written informed consent dated and signed by the patient

Exclusion Criteria:

* All other breast cancers than those described in inclusion criteria, in particular inflammatory and/or neglected (T4b or T4d) forms.
* Patient presenting with plurifocal tumors, multicentric tumor, bilateral tumor.
* Grade I well differentiated tumor.
* HER2 neu 3 + (ICH or FISH or CISH) tumor.
* Non measurable lesion, in the two diameters, whatever radiological methods used.
* Patient presenting microcalcifications for which breast conservation is not possible.
* Patient already operated for breast cancer or having had primary axillar node dissection.
* Patient having antecedent of other cancer, exception for in situ uterine cervix or basocellular skin cancer, considered as healed.
* Patient presenting another pathology considered as incompatible with patient inclusion in the study
* Patient should not receive treatment with any other investigational drug and should not participate to another clinical study in a delay < 30 days or should not be pre-treated by cytostatic chemotherapy.
* Antecedents of allergy to polysorbate 80.
* Patient who is pregnant or lactating and not using effective contraceptive method.
* Any psychological, familial, sociological or geographical condition that may potentially hamper compliance with the study protocol and follow up schedule, assessed with the patient prior to registration in the trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2007-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Improvement of complete pathological response rate at surgery after 6 chemotherapy cycles | after 6 cycles of chemotherapy

SECONDARY OUTCOMES:
Tolerance according to NCI-CTC criteria | after each cycle of chemotherapy
Objective clinical, echographic, mammographic responses after 6 cycles | after every 2 cycles of chemotherapy treatment
Breast conservation rate | at surgery
Study of biological predictive factors of chemosensitivity and resistance by immunological and molecular biology techniques) | before receive chemotherapy
Overall and relapse-free survivals | 5 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chollet, Pr, Study Chair — Centre Jean Perrin
Locations (6):
- France (6):
  - Hospital center, Brive-la-Gaillarde
  - Centre Jean Perrin, Clermont-Ferrand
  - University Hospital La Tronche, Grenoble
  - Edouard Herriot University Hospital, Lyon
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Background] Roché H, Fumoleau P, Spielman M et al. Breast Cancer Res Treat. 2004;88(suppl1):S16. Abstract 27
- [Background] Mouret-Reynier MA, Abrial CJ, Ferriere JP, Amat S, Cure HD, Kwiatkowski FG, Feillel VA, Lebouedec G, Penault-Llorca FM, Chollet PJ. Neoadjuvant FEC 100 for operable breast cancer: eight-year experience at Centre Jean Perrin. Clin Breast Cancer. 2004 Oct;5(4):303-7. doi: 10.3816/cbc.2004.n.035. PMID 15507178
- [Derived] Wang-Lopez Q, Mouret-Reynier MA, Savoye AM, Abrial C, Kwiatkowski F, Garbar C, DuBray-Longeras P, Eymard JC, Lebouedec G, Vanpraagh I, Penault-Llorca F, Chollet P, Cure H. Is it important to adapt neoadjuvant chemotherapy to the visible clinical response? An open randomized phase II study comparing response-guided and standard treatments in HER2-negative operable breast cancer. Oncologist. 2015 Mar;20(3):243-4. doi: 10.1634/theoncologist.2014-0400. Epub 2015 Jan 30. PMID 25637380